CLINICAL TRIAL: NCT02714829
Title: Clinical Study to Evaluate Efficacy and Safety of "Inject BMP(Beta-TCP Containing rhBMP-2)" for Socket Preservation After Extraction of a Single-rooted Tooth: A Randomized, Outcomes Assessor-Blinded, Multi-center, Prospective Trial.
Brief Title: Clinical Study of Injectable Ceramics Bone Graft Substitute Containing rhBMP-2
Acronym: rhBMP-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioAlpha Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ExcelOS 14-01
Record Dates: First submitted 2016-03-08; First posted 2016-03-22 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Alveolar Bone Preservation; Bone Graft
Keywords: Injectable Ceramics Bone Graft Substitute Containing rhBMP-2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inject BMP (Experimental): ExcelOS-inject containing rhBMP-2
  Interventions: Device: Inject BMP
- ExcelOS-inject (Active Comparator): ExcelOS-inject without rhBMP-2
  Interventions: Device: ExcelOS-inject

INTERVENTIONS:
Device: Inject BMP — Injection of ExcelOS-inject(beta-TCP) containing rhBMP-2.
  Arms: Inject BMP
Device: ExcelOS-inject — Injection of ExcelOS-inject(beta-TCP) without rhBMP-2.
  Arms: ExcelOS-inject

SUMMARY:
This is a prospective, outcomes assessor-blinded, randomized study to evaluate the efficacy and safety of "Inject BMP(Injectable Ceramics Bone Graft Substitute Containing rhBMP-2)" for socket preservation after extraction of a single-rooted tooth, compared to ExcelOS-inject(Injectable Ceramics Bone Graft Substitute).

DETAILED DESCRIPTION:
Inject BMP is Injectable Ceramics Bone Graft Substitute(ExcelOS-inject) containing rhBMP-2. Recombinant human Bone morphogenetic protein 2 (rhBMP-2) stimulates the production of bone.

ELIGIBILITY:
Inclusion Criteria:

* Persons without periodontal disease

Exclusion Criteria:

* Women who are pregnant or plan to be pregnant within study period

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
compared the changed height and standard height by computed tomography. | at 12 weeks after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Soon Jung Hwang, Ph.D, Principal Investigator — Seoul National University Dental Hospital; Jong-Rak Hong, Ph.D, Principal Investigator — Samsung Medical Center; Hee-Kyun Oh, Ph.D, Principal Investigator — Chonnam National University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Han JJ, Chang AR, Ahn J, Jung S, Hong J, Oh HK, Hwang SJ. Efficacy and safety of rhBMP/beta-TCP in alveolar ridge preservation: a multicenter, randomized, open-label, comparative, investigator-blinded clinical trial. Maxillofac Plast Reconstr Surg. 2021 Dec 20;43(1):42. doi: 10.1186/s40902-021-00328-0. PMID 34928477